CLINICAL TRIAL: NCT04893161
Title: A Model to Early Predict the Response of Belimumab Treatment in the Patients With Systemic Lupus Erythematosus
Brief Title: A Model About the Response of Belimumab in SLE
Acronym: MRBS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2020LSK-278
Record Dates: First submitted 2021-05-16; First posted 2021-05-19 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-01

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab

STUDY DESIGN:
Intervention Model Description: All patients with SLE will be enrolled in one year and administrated belimumab 10mg/kg intravenous infusion over 1 hour on days 0, 14, and 28, and every 28 days through week 48.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- belimumab (Other): All patients with SLE receive belimumab 10mg/kg intravenous infusion over 1 hour on days 0, 14, and 28, and every 28 days through week 48. The patients who had SRI-4 response at week 48 were divided into response group and the patients without SRI-4 response at week 48 were divided into no response group.
  Interventions: Drug: Belimumab

INTERVENTIONS:
Drug: Belimumab — All patients with SLE will be enrolled in one year and administrated belimumab 10mg/kg intravenous infusion over 1 hour on days 0, 14, and 28, and every 28 days through week 48.
  Other Names: The standard care

SUMMARY:
A prospective, single-center cohort study aims to determine a predictive model of the response of belimumab at Week 48.

DETAILED DESCRIPTION:
Preamble:

Belimumab is an inhibitor of B cell activating factor (BAFF) that has been developed as an agent for the treatment of patients with systemic lupus erythematosus (SLE).

In July 2019, belimumab was approved for marketing in China. The belimumab treatment has been proved to reduce the level of autoantibodies and control disease activity in the patients with SLE. The response rate of SLE Responder Index-4 (SRI-4) is approximately 50% in the BLISS-52 and BLISS-76 phase III clinical trials. The goal of this study is to establish a predictive model (including immune marker, inflammatory biomarker and clinical factor) to early estimate the response of belimumab treatment.

Objectives:

Primary objective: in the patients with SLE, an early predictive model of the response of belimumab treatment will be estimated.

Secondary objectives:

In subjects with SLE receiving belimumab treatment, to assess the effect of belimumab on:

The clinical improvement; The serological variables improvemen. The inflammatory biomarkers improvemen. The quality of life. The dosage of prednisone. The kinetics of B cell phenotype. The function of non-switched memory B cells. The association between the immune, inflammatory and clinical markers and the response of belimumab.

The mechanism of BAFF inhibition on the survival and selection of SLE non-switched memory B cells.

The recovering of immune checkpoint in non-switched memory B cells from the view of BCR mutation.

The rates of adverse events.

Overview of study design:

This is a prospective, single-center cohort study to estimate a predictive model of the response of belimumab. All patients with SLE receive belimumab 10mg/kg intravenous infusion over 1 hour on days 0, 14, and 28, and every 28 days through week 48. All patients are evaluated at week 0, 2, 4, 8, 12, 24, 36, and 48. The immune markers, inflammatory biomarkers, clinical markers and safety data are assessed following belimumab treatment.

Study population:

Men or women with SLE who have active (according to SLEDAI-2K) and refractory SLE manifestations. SLE manifestations are deﬁned as refractory in case of drug intolerance, unresponsiveness, or disease relapse in patients treated with corticosteroids, antimalarials, and/or immunosuppressants. Patients with renal disease were considered as refractory when they had a persistence of 24 hours proteinuria > 1 g after at least 1 year from the start of the initial therapy or when they experienced a renal ﬂare (24 hours proteinuria > 1 g in case of previous complete response or doubling 24 hours proteinuria in other cases) during the subsequent therapy.

ELIGIBILITY:
Inclusion Criteria:

* Fulfillment of the 1997 American College of Rheumatology (ACR) revised criteria for SLE;
* Aged more than 18 years;
* Active (according to SLEDAI-2K) and refractory SLE manifestations. SLE manifestations are deﬁned as refractory in case of drug intolerance, unresponsiveness, or disease relapse in patients treated with corticosteroids, antimalarials, and/or immunosuppressants. Patients with renal disease were considered as refractory when they had a persistence of 24 hours proteinuria > 1 g after at least 1 year from the start of the initial therapy or when they experienced a renal ﬂare (24 hours proteinuria > 1 g in case of previous complete response or doubling 24 hours proteinuria in other cases) during the subsequent therapy.

Exclusion Criteria:

* Have a history of malignant neoplasm within the last 5 years except basal cell or squamous cell carcinoma of the skin treated with local resection only or carcinoma in situ of the uterine cervix treated locally and with no evidence of metastatic disease for 3 years;
* Have evidence of serious suicide risk including any history of suicidal behaviour in the last 6 months and/or any suicidal ideation in the last 2 months or who in the investigator's judgment, poses a significant suicide risk;
* Have a history of a primary immunodeficiency;
* Have a significant IgG deficiency (IgG level < 400 mg/dL);
* Have an IgA deficiency (IgA level < 10 mg/dL)
* Have cyclophosphamide or rituximab treatment.
* Infection history:

Currently on any suppressive therapy for a chronic infection (such as tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster and atypical mycobacteria) Hospitalization for treatment of infection within 60 days of Day 0; Use of parenteral (IV or IM) antibiotics (anti-bacterial, antiviral, anti-fungal, or anti-parasitic agents) within 60 days of Day 0.

* Have current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence within 365 days prior to Day 0;
* Have a historically positive HIV test or test positive at screening for HIV;
* Hepatitis status:

Serologic evidence of current or past Hepatitis B (HB) infection based on the results of testing for HBsAg and HBcAb as follows:

Patients positive for HBsAg or HBcAb are excluded Positive test for Hepatitis C antibody

* Have a history of an anaphylactic reaction to parenteral administration of contrast agents, human or murine proteins or monoclonal antibodies;
* Have any other clinically significant abnormal laboratory value in the opinion of the investigator;
* Have any intercurrent significant medical or psychiatric illness that the investigator considers would make the candidate unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Establishment of predictive model to assess the SRI response rate. | at week 48
  An SRI response is defined as a ≥ 4-point reduction in SELENA-SLEDAI score, no new BILAG A organ domain score and no more than 1 new BILAG B score, and no worsening (increase < 0.3) in PGA score versus baseline.

SECONDARY OUTCOMES:
The SRI-4 response rate | at week 48
  An SRI response is defined as a ≥ 4-point reduction in SELENA-SLEDAI score, no new BILAG A organ domain score and no more than 1 new BILAG B score, and no worsening (increase < 0.3) in PGA score versus baseline.
The rate of adverse events | week 0 to week 48
  all adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Lan He, Dr., Study Chair — First Affiliated Hospital Xi'an Jiaotong University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang J, Ju B, Zhu L, Li H, Luo J, Zhang J, Hu N, Mo L, Wang Y, Pan Y, Huang J, Lv X, Pu D, Hao Z, He L, Li Y. The rapid inhibition of B-cell activation markers by belimumab was associated with disease control in systemic lupus erythematosus patients. Front Pharmacol. 2023 Feb 16;14:1080730. doi: 10.3389/fphar.2023.1080730. eCollection 2023. PMID 36873989